CLINICAL TRIAL: NCT06998771
Title: A Phase II Trial to Evaluate the Safety and Efficacy of JSKN003 Combination Therapy as First-line Treatment in HER2-positive Unresectable Locally Advanced or Metastatic Gastric Cancer or Resectable Gastric Cancer
Brief Title: JSKN003 Combined Treatment of HER2-positive Gastric Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JSKN003-003
Record Dates: First submitted 2025-05-12; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: HER2-positive Gastric Cancer
MeSH Terms: interventions — Capecitabine; Oxaliplatin; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Combination of JSKN003 and capecitabine with or without enlonstobart (Experimental)
  Interventions: Drug: JSKN003; Drug: Capecitabine; Drug: Enlonstobart
- Combination of JSKN003, capecitabine and KN026 with or without enlonstobart (Experimental)
  Interventions: Drug: JSKN003; Drug: KN026; Drug: Capecitabine; Drug: Enlonstobart
- Combination of JSKN003, capecitabine and oxaliplatin with or without enlonstobart (Experimental)
  Interventions: Drug: JSKN003; Drug: Capecitabine; Drug: Enlonstobart; Drug: Oxaliplatin
- Combination of trastuzumab, capecitabine and oxaliplatin with or without pembolizumab (Experimental)
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin; Drug: Trastuzumab; Drug: Pembolizumab

INTERVENTIONS:
Drug: JSKN003 — JSKN003 is administered by intravenous infusion.
  Arms: Combination of JSKN003 and capecitabine with or without enlonstobart; Combination of JSKN003, capecitabine and KN026 with or without enlonstobart; Combination of JSKN003, capecitabine and oxaliplatin with or without enlonstobart
Drug: KN026 — KN026 is administered by intravenous infusion.
  Arms: Combination of JSKN003, capecitabine and KN026 with or without enlonstobart
Drug: Capecitabine — Capecitabine is for oral administration.
Drug: Enlonstobart — Enlonstobart is administered by intravenous infusion.
  Arms: Combination of JSKN003 and capecitabine with or without enlonstobart; Combination of JSKN003, capecitabine and KN026 with or without enlonstobart; Combination of JSKN003, capecitabine and oxaliplatin with or without enlonstobart
Drug: Oxaliplatin — Oxaliplatin is administered by intravenous infusion.
  Arms: Combination of JSKN003, capecitabine and oxaliplatin with or without enlonstobart; Combination of trastuzumab, capecitabine and oxaliplatin with or without pembolizumab
Drug: Trastuzumab — Trastuzumab is administered by intravenous infusion.
  Arms: Combination of trastuzumab, capecitabine and oxaliplatin with or without pembolizumab
Drug: Pembolizumab — Pembolizumab is administered by intravenous infusion.
  Arms: Combination of trastuzumab, capecitabine and oxaliplatin with or without pembolizumab

SUMMARY:
This study is designed to evaluate the safety and efficacy of JSKN003 combination therapy as first-line treatment in HER2-positive unresectable locally advanced or metastatic gastric cancer or resectable gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years old.
* Histologically or cytologically confirmed diagnosis of gastric cancer.
* The first-line population enrolls participants with HER2-positive unresectable locally advanced or metastatic gastric cancer who had not received systemic treatment, and Perioperative population enrolls participants with HER2-positive resectable gastric cancer who had not received treatment.
* HER2-positive (defined as IHC3+ or IHC 2+/FISH +).
* The first-line population: presence of at least 1 measurable lesion per RECIST 1.1. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* ECOG PS of 0 - 1.
* Expected survival ≥ 3 months.
* Participants with adequate organ functions.
* Female and male patients of childbearing age agree to take adequate contraceptive measures during and upon completion of the study for 7 months after the last dose. Female participants of childbearing age must have a negative blood pregnancy test within 7 days before the first dose or randomization.
* Voluntarily agree to participate in the study and sign the informed consent.

Exclusion Criteria:

* Has received anti-tumor treatment such as systemic chemotherapy or other trial interventions within 28 days, or immunotherapy (e.g. interleukin, interferon, thymospipeptide, etc.), hormone therapy or targeted therapy within 14 days or 5 half-life (whichever is shorter) before the first dose or randomization.
* Has previously been treated with an anti-HER2 ADC loaded with topoisomerase I inhibitors.
* Participants with brain metastasis or spinal cord compression at screening (except for completed local treatment and discontinued glucocorticoids for at least 4 weeks before the first dose or randomization , and stable central nervous system imaging and brain metastasis symptoms for at least 4 weeks).
* Participants with PD-L1 CPS ≥1, who are receiving long-term immunotherapy (e.g., cyclosporine) or require daily systemic steroid therapy (e.g., >20 mg prednisone or equivalent), except those who treated with local glucocorticoids using nasal spray, inhalation, or other pathways.
* Participants with PD-L1CPS ≥1, who have an active autoimmune disease or have a history of autoimmune disease 2 years before the first dose or randomization and still require systemic treatment. However, participant with the following diseases is allowed to enroll: well-controlled type I diabetes, well-controlled hypothyroidism that requires hormone replacement therapy, skin diseases that do not require systemic treatment (such as vitiligo, psoriasis, or hair loss), or participant who is expected to not recur without external triggers.
* Participate in another clinical trial, unless it is an observational (non-intervention) clinical trial or is in the follow-up period of an intervention trial.
* Participants who have undergone major surgery or had invasive intervention within 28 days before the first dose or randomization. Or those who plan to undergo systematic or local tumor resection during the trial (Perioperative cohort does not apply).
* Any Chinese patent medicine with anti-cancer activity approved by the National Drug Administration (regardless of cancer type) has been used within 14 days before the first dose or randomization.
* Has a history of severe hypersensitivity reactions to either the drug substances or inactive ingredients in the drug product.
* Active bacterial, fungal or viral infection before the first dose or randomization. Participant who has recieved preventive infection treatment but has no clinical manifestations before the first dose or randomization could be considered to enroll.
* Has a history of immunodeficiency, including HIV-positive.
* Active hepatitis B or C infection. Participant with positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) need to test Hepatitis B virus DeoxyriboNucleic Acid (HBV-DNA), and HBV-DNA is higher than 500 IU/mL (or 2500 copies/ml) or upper limit of normal (UNL) (whichever is lower) ; Participants with positive for hepatitis C (HCV) antibody and whose Hepatitis C virus Ribonucleic Acid (HCV-RNA) is higher than 1000 copies/ml or UNL (whichever is lower).
* Has a history of tuberculosis treatment within 2 years before the first dose or randomization.
* Has activity or a history of interstitial lung disease at any stage and/or pulmonary function injury, a history of interstitial pneumonia requiring hormone therapy, or the imaging cannot rule out suspected interstitial lung disease/pneumonia at screening.
* Known to have low activity or lack of dihydropyrimidine dehydrogenase (DPD).
* Participants with peripheral neuropathy of grade > 1.
* Participants with clinically significant gastrointestinal diseases including but not limited to severe liver diseases, ulcerative colitis, inflammatory bowel disease and other gastrointestinal diseases 28 days before the first dose or randomization.
* Has a history of severe cardiovascular disease.
* History of any other malignant tumors within 5 years before the first dose or randomization.
* Live vaccination within 28 days before the first dose or randomization. Note: Seasonal influenza vaccine is a broadly inactivated vaccine and is allowed to be used;
* Unable to swallow orally, or there are conditions that have been judged by researchers to seriously affect gastrointestinal absorption (such as severe Crohn's disease, malabsorption syndrome, etc.).
* Pregnant or breastfeeding women.
* Otherwise considered inappropriate for the study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) of the first-line population | Frame: Up to approximately 5 years
Incidence and severity of TEAE and SAE of the first-line population | Up to approximately 5 years
pCR rate after neoadjuvant therapy of perioperative population | Up to approximately 5 years

SECONDARY OUTCOMES:
Disease Control Rate (DCR) of the first-line population | Up to approximately 5 years
Duration of Response (DoR) of the first-line population | Up to approximately 5 years
Progression-free survival (PFS) of the first-line populations | Up to approximately 5 years
Major pathological response (MPR) rate of perioperative population | Up to approximately 5 years
R0 rate of perioperative population | Up to approximately 5 years
Event-free survival (EFS) of perioperative population | Up to approximately 5 years
Overall Survival (OS) | Up to approximately 5 years
Incidence and severity of AE | Up to approximately 5 years
Blood concentration of JSKN003 | Up to approximately 2 years
Blood concentration of total antibodies for JSKN003 | Up to approximately 2 years
Blood concentration of free toxins for JSKN003 | Up to approximately 2 years
Serum concentration of KN026 | Up to approximately 2 years
Serum concentration of Enlonstobart; | Up to approximately 2 years
Anti-drug antibodies (ADA) related to JSKN003 | Up to approximately 2 years
Title: ADA related to KN026 | Up to approximately 2 years
ADA related to Enlonstobart | Up to approximately 2 years